CLINICAL TRIAL: NCT00738387
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Multi-center Study of ASA404 in Combination With Docetaxel in Second-line Treatment of Patients With Locally Advanced or Metastatic (Stage IIIb/IV) Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of ASA404 or Placebo in Combination With Docetaxel in Second-line Treatment for (Stage IIIb/IV) Non-small Cell Lung Cancer
Acronym: ATTRACT-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASA404A2302; EUDRACT number: 2008-002309-38
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2012-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Tumor vascular disrupting agent; VDA; ASA404; non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vadimezan; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ASA404 + docetaxel (Experimental): 1800 mg/m2 of ASA404 intravenous (IV) on day 1 of each 21 day cycle
  75 mg/m2 of docetaxel intravenous (IV) an hour for 1st 6 cycles; cycle: every 21 days
  Interventions: Drug: ASA404; Drug: docetaxel
- Placebo + docetaxel (Placebo Comparator): Placebo i.v. on day 1 of each 21 day cycle
  75 mg/m2 of docetaxel intravenous (IV) an hour for 1st 6 cycles; cycle: every 21 days
  Interventions: Drug: Placebo; Drug: docetaxel

INTERVENTIONS:
Drug: ASA404 — 1800 mg/m2 of ASA404 i.v. on day 1 of each 21 day cycle
  Arms: ASA404 + docetaxel
Drug: Placebo — Placebo i.v. on day 1 of each 21 day cycle
  Arms: Placebo + docetaxel
Drug: docetaxel — 75 mg/m2 of docetaxel intravenous (IV) an hour for 1st 6 cycles; cycle: every 21 days

SUMMARY:
The purpose of this study is to determine if adding ASA404 to docetaxel chemotherapy makes the cancer treatment more effective in patients with locally advanced or metastatic non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell carcinoma of the lung of all histologies. (Histological or cytological specimens must be collected via surgical biopsy, brushing, washing or core needle aspiration of a defined lesion. Sputum cytology is not acceptable.)
2. Patients who have progressed while on or following a first-line chemotherapy regimen for Stage IIIb disease (malignant pleural effusion or pericardial effusion that have been confirmed cytologically) or Stage IV disease. Patients who have received bevacizumab and/or EGFR inhibitors in first-line will be eligible
3. Age ≥ 18 years old
4. WHO Performance Status of 0-2
5. Not applicable per amendment#2
6. Central laboratory values within the range, as defined below, within 2 weeks of randomization:

   * Absolute neutrophils count (ANC) ≥ 2.0 x 109/L
   * Platelets ≥ 100 x109/L
   * Hemoglobin ≥ 10 g/dL
   * Serum creatinine ≤ 1.5 x ULN
   * Serum bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN (≤5 x ULN if liver metastases)
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 x ULN
   * Electrolyte values (sodium, potassium, calcium, magnesium) within ≥1 x LLN and ≤1 x ULN. Patients with corrected electrolyte values are eligible
   * Females of child-bearing potential must have negative serum pregnancy test (confirmation of negative urine pregnancy test within 72 hours prior to initial dosing). Any female presenting with a positive or borderline pregnancy test may undergo a gynecological exam and ultra sound to rule out pregnancy and if found to be negative may be included in the trial.
7. Life expectancy ≥ 12 weeks
8. Written informed consent obtained according to local guidelines

Exclusion Criteria:

1. Patients having CNS metastases (patients having any clinical signs of CNS metastases must have a CT or MRI of the brain performed to rule out CNS metastases in order to be eligible for study participation. Patients who have had brain metastases surgically removed or irradiated with no residual disease confirmed by imaging are allowed).
2. Patients with concurrent malignancy, or history or prior malignancy within the past two years, except for basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, treated early stage (T1a) prostate cancer or treated early stage (DCIS or LCIS) breast cancer.
3. Radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered from all acute radiotherapy-related toxicities.
4. Major surgery must be completed 4 weeks prior to starting study treatment. Major surgery is defined at the investigator's discretion. Insertion of a vascular access device is not considered major or minor surgery. Patients must have recovered from all acute surgery-related complications.
5. Treatment with all prior anticancer therapies ≤ 3 weeks prior to randomization (≤ 6 weeks for bevacizumab, mitomycin and nitrosoureas)
6. Concurrent use of other investigational agents and patients who have received investigational agents ≤ 4 weeks prior to randomization
7. Prior treatment with docetaxel for NSCLC in the locally advanced or metastatic first-line setting
8. Prior treatment with VDAs or tumor - VDAs
9. Any medical condition resulting in ≥ CTC grade 2 dyspnea
10. Patients with systolic BP > 160 mm Hg and/or diastolic BP > 90 mm Hg while on medication for hypertension
11. Patients with recent hemoptysis associated with NSCLC (>1 teaspoon in a single episode within 4 weeks)
12. Patients with any one of the following:

    * Patients with long QT syndrome
    * Patients with a Baseline 12-lead ECG QTcF of > 450 msec for men or >470 msec for women using the Fridericia [QTcF formula] measurement determined per central ECG evaluation report
    * Congestive heart failure (NY Heart Association class III or IV)
    * Patients with a myocardial infarction within 12 months of starting study treatment or with implanted cardiac pacemaker
    * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
    * History of poorly-controlled hypertension or poor compliance with anti-hypertensive regimen
    * History of a sustained ventricular tachycardia
    * Presence of atrial tachycardia (e.g., atrial fibrillation, atrial flutter, multifocal atrial tachycardia, supraventricular tachycardia) if not effectively rate-controlled
    * History of ventricular fibrillation or Torsades de Pointes (TdP)
    * Right bundle branch block (RBBB) and either left anterior hemiblock or left posterior hemiblock (bifasicular block)
    * Bradycardia defined as heart rate <50 beats per minute
    * [For China only: Patients older than 70 years with evidence of myocardial ischemia by coronary artery angiography or cardiac radionucleotide imaging examination]
    * [For China only: Patients with LVEF <=40%]
    * Any clinically significant cardiac abnormality as assessed by the investigator
13. Patients who are currently receiving treatment with any medications that have the potential to prolong QT interval or are known to have a risk of causing Torsades de Pointes (See Section 6.8.5.1 and Appendix 2) which cannot be either safely discontinued or switched to a different medication prior to starting study drug administration must be discussed with and approved by the Novartis Global Clinical team prior to randomization.
14. Known allergy or hypersensitivity to docetaxel or drugs formulated with polysorbate 80
15. Peripheral sensory neuropathy with functional impairment (CTC grade 2 neuropathy, regardless of causality)
16. Pregnant or breast feeding females

    • Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml)
17. Women of child bearing potential or sexually active males, unwilling or unable to use the required highly effective method(s) of contraception for both sexes while receiving treatment and for at least 6 months after the discontinuation of study treatment. (Adequate forms of contraception include IUD, oral or depot contraceptive or the barrier method plus spermicide.)

    • Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions while taking docetaxel and therefore are not considered effective contraceptive methods for this study when used as a single agent. Therefore, it is highly recommended that a concomitant barrier method be used with oral, implantable, or injectable contraceptives. The investigator shall counsel the patient accordingly. Women of childbearing potential must have a negative pregnancy test (serum or urine) 72 hours prior to administration of study treatment. For a list of substrates of human liver microsomal P450 enzymes, visit website (http://medicine.iupui.edu/flockhart/)
18. Concurrent severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, chronic renal disease, chronic liver disease, confirmed diagnosis of HIV infection or active uncontrolled infection).
19. Significant neurologic or psychiatric disorder which could compromise participation in the study
20. Patient unwilling or unable to comply with the protocol
21. Patients receiving full-dose therapeutic oral or parenteral anticoagulation are ineligible. Patients receiving thrombolytic therapy within 10 days of starting are also ineligible.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | Every 6 weeks from study treatment discontinuation until death or loss to follow-up

SECONDARY OUTCOMES:
Progression free survival | Every 6 weeks from study treatment discontinuation until documented PD, death or loss to follow-up
Overall response rate | Every 42 days (=/- 7 days) from date of randomization until PD
Quality of life | At every odd cycle and at end of treatment
Biomarker assessments | 1 hr post-study drug at cycles 1, 2, 4, 6 and End of Treatment
Pharmacokinetic assessments | 1 hr post-study drug, optional 3-5 hr post-study drug at cycles 1, 2, 3, 4, 5 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (162):
- United States (88):
  - Oncology Specialist, P.c., Huntsville, Alabama
  - Arizona Oncology, Tucson, Arizona
  - Highlands Oncology Group, Bentonville, Arkansas
  - Central Hematology Oncology Medical Group, Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Compassionate Cancer Care Medical Group, Corona, California
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Beaver Medical Group, L.P., Highland, California
  - Scripps Clinic, La Jolla, California
  - University of Southern Californa, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - University of California Irvine Medical Center, Orange, California
  - Ventura County Hematology/Oncology Specialists, Oxnard, California
  - Palo Alto Medical Foundation - Camino Div., Palo Alto, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Loma Linda Oncology Medical Group, Inc., Redlands, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - California Pacific Medical Research Institute, San Francisco, California
  - University of California - SF, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Advanced Medical Specialties, Miami, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Cancer Centers of Florida, PA, Orlando, Florida
  - Hematology/Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Suburban Hematology-Oncology, Lawrenceville, Georgia
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Comprehensive Cancer Program, Harvey, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - OSF Center for Cancer Care, Rockford, Illinois
  - Loyola Cancer Care and Research Center, Winfield, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Kansas City Cancer care, Southwest, Overland Park, Kansas
  - University of Kansas Medical Center, Westwood, Kansas
  - Cancer Center of Texas, Wichita, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Western Kentucky Hematology & Oncology, Paducah, Kentucky
  - Harry & Jeannette Weinberg Cancer Institute, Baltimore, Maryland
  - Missouri Cancer Associates, Columbia, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Advanced Oncology Associates, Armonk, New York
  - Arena Oncology Associates, P.C., Lake Success, New York
  - NY Oncology/Hematology - Latham, Latham, New York
  - Winthrop Hematology/Oncology, Mineola, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cancer Center of North Carolina, Raleigh, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Hematology Oncology Consultants, Inc., Columbus, Ohio
  - Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Kaiser Permanante, Northwest Region, Portland, Oregon
  - St. Luke's Hospital & Healtth Network, Bethlehem, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Cancer center - Abilene, Abilene, Texas
  - Texas Oncology - Arlington South, Arlington, Texas
  - Mamie McFadden Ward Cancer Ctr, Texas Oncology, Beaumont, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology at Presbyterian Hospital, Dallas, Texas
  - Methodist Charlton Cancer Center, Dallas, Texas
  - UT Southwester Med Ctr at Dallas, Dallas, Texas
  - Texas Cancer Center - Denton, Denton, Texas
  - Longview Cancer Center, Longview, Texas
  - Texas Oncology - Allison Cancer Center, Midland, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Texas Oncology Cancer Care Center & Research Center, Waco, Texas
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Fred Hutchinson Cancer Reseach Center, Seattle, Washington
  - Puget Sound Cancer Center, Seattle, Washington
  - Evergreen Hematology and Oncology, Spokane, Washington
  - MultiCare Health System, Tacoma, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
- Belgium (8):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Arlon
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
- Canada (9):
  - Novartis Investigative Site, Edmonton
  - Novartis Investigative Site, Greenfield Park
  - Novartis Investigative Site, Laval
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Toronto
  - Novartis Investigative Site, Trois-Rivières
  - Novartis Investigative Site, Vancouver
  - Novartis Investigative Site, Weston
  - Novartis Investigative Site, Winnepeg
- France (11):
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, La Chaussée-Saint-Victor
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (19):
  - Novartis Investigative site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Eschweiler
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Güstrow
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hemer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Ulm
- Hungary (5):
  - Novartis Investigative site, Deszk
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Törökbálint
  - Novartis Investigative Site, Zalaegerszeg-Pozva
- Italy (13):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Cosenza
  - Novartis Investigative Site, Cremona
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Mirano
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Sassari
  - Novartis InvestigativeSite, Udine
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lonza
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
- Spain (3):
  - Novartis Investigative Site, Mataró
  - Novartis investigative Site, Sabadell
  - Novartis Investigative Site, Santander
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative site, Sankt Gallen

REFERENCES:
- See also: Results for CASA404A2302 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4927